CLINICAL TRIAL: NCT03738631
Title: Association of Cardiac Biomarker Elevation After Marathon Running and Coronary Atherosclerosis - the MaraCat Study
Brief Title: Cardiac Biomarkers After Marathon Running and Coronary Atherosclerosis
Acronym: MaraCat
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor, Turku University Hospital
Other Study IDs: T171/2018
Record Dates: First submitted 2018-09-21; First posted 2018-11-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Under 35 years
- Over 44 years

SUMMARY:
This study evaluates cardiac biomarkers and their association to coronary artery disease in marathon runners.

DETAILED DESCRIPTION:
The MaraCat study is an observational prospective study evaluating the association between cardiac biomarkers and coronary artery disease in 43 runners participating in the 2018 Paavo Nurmi Marathon. The study participants were recruited according to two age criteria - under 35 years and over 44 years of age. Comprehensive laboratory samples were collected immediately after the run, while the control workup was done in a separate visit with no significant physical excercise in the preceding two weeks. In the under 35 years -group, the control workup included an echocardiography, ecg and blood samples. In the over 44 years group, the control studies included coronary CT, echocardiography, ecg and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Age under 35 years or over 44 years
* Participant of Paavo Nurmi Marathon 2018
* Informed consent signed

Exclusion Criteria:

* No informed consent
* existing coronary artery disease

Ages: 35 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male participants of the Paavo Nurmi Marathon 2018
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Cardiac Troponin-T level after marathon | 0-30minutes after finishing the Paavo Nurmi Marathon
  Cardiac troponin-T levels (ng/L), [electrochemiluminescence (ECLIA) method]
Association Cardiac troponin-T level and coronary CT findings | Cardiac Troponin-T 0-30 minutes after finishing the Paavo Nurmi Marathon. Control Troponin-T levels and coronary CT angiography at control visit (>30days after marathon).
  Cardiac troponin-T levels (ng/L), [electrochemiluminescence (ECLIA) method]

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Heart Center, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided